CLINICAL TRIAL: NCT02125045
Title: Medium Term Effect of Sublingual L-glutathione (L-GSH) Supplementation on Flow Mediated Dilation and Oxidative Stress Markers in Male Subjects With Smoking Habit and/or Arterial Hypertension
Brief Title: Sublingual L-GSH Supplementation in Male Subjects With Smoking Habit and/or Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 215_062013
Record Dates: First submitted 2013-11-26; First posted 2014-04-29 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Health Subjects With Cardiovascular Risk Factors
Keywords: GSH; cardiovascular risk factors; endothelial dysfunction; oxidative stress

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-GSH (Experimental): Glutathione 100 mg tablets twice a day
  Interventions: Dietary Supplement: L-GSH
- Placebo (Placebo Comparator): Matching placebo will be administered for 4 weeks in a double blind fashion.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-GSH — Reduced glutathione is formed by cysteine, glycine and glutamate. It enters into the detoxification processes of endogenous products, such as peroxides which are the final pathway of many reactions caused by cardiovascular risk factors. It also acts on the exogenous compounds, such as pollutants, heavy metals and some drugs.
  Arms: L-GSH
Dietary Supplement: Placebo — Placebo will be prepared using the same excipients of the dietary supplement without active substance.
  Arms: Placebo

SUMMARY:
Background. The antioxidant systems are the main endogenous defense against free radicals, and glutathione seems to play an important role in this mechanism. Reduced glutathione enters into the detoxification processes of endogenous products, such as hydro- and lipoperoxides and exogenous compounds such as pollutants, heavy metals and some drugs. Changes in GSH homeostasis have been implicated in the etiology and progression of several diseases. Supplementation of GSH may improve the endogenous antioxidant defense and may contribute to decrease of oxidants tissue damage a pathophysiologic mechanism of many acute and chronic diseases.

However, the efficacy of GSH treatment seems to be closely related to the degree of its absorption and to the increase of its concentrations in plasma and cells. Previous studies of oral GSH administration in healthy volunteers or in patients failed to find any effect in terms of oxidative stress reduction and/or disease improvement because the GSH is quickly catabolized by gastrointestinal tract. We have recently observed (preliminary data) that a new sublingual formulation of L-GSH (OXITION), produced by PH&T S.r.l., is able to increase erythrocyte and plasma GSH levels in healthy volunteers bypassing gastrointestinal barrier.

Objectives. The primary study objective is to determine whether medium term (4 weeks) of sublingual L-GSH supplementation to a population with smoking habit and/or arterial hypertension may result in improved endothelial function as assessed by the flow mediated dilation (FMD) technique versus placebo. FMD is a surrogate end point validated in the literature as prognostic predictor for major cardiovascular events in patients with endothelial dysfunction. Secondary study objectives are to determine differences between the 2 treatment in terms of oxidative stress markers.

Methods. This is a phase 3, double-blind, randomized, placebo-controlled, cross-over study performed in only one centre. Sixteen male subjects, aged ≥ 40 and ≤ 60 years, with smoking habit and/or hypertension defined as arterial blood pressure ≥ 140 and/or 90 mmHg or in anti-hypertensive treatment, will be enrolled and randomized to receive sublingual L-GSH (100 mg twice a day) or placebo according to a double-blind cross-over design for 4 weeks with a 3-week wash-out period between the two treatments. Baseline and at the end of each treatment period, FMD assessment and blood samples collection for routine (creatinine, urea, AST, ALT GGT, total cholesterol, HDL, LDL, triglycerides, fasting glucose) and specific (aminothiols, nitrotyrosine, malondialdehyde, 8-hydroxy-deoxyguanine) biochemical determination will be performed.

DETAILED DESCRIPTION:
The strategies to prevent cardiovascular diseases play a prominent role in the guidelines of different scientific societies. Risk factors lead to several biological reactions within the cell in terms of pathophysiology, and thus of response to the homeostasis alteration. It is known that both smoking habit and hypertension alters endothelial functions through direct oxidative damage to endothelial cells, decrease in nitric oxide availability, and affects the mobilization of endothelial progenitor cells from the bone marrow.

Several studies have identified this response in the activation of mechanism that prevent the formation of oxidizing species, detoxifying any dangerous products. The antioxidant systems are, thus, the main endogenous defense against free radicals, and glutathione seems to play an important role in this mechanism. Reduced glutathione (GSH), formed by cysteine, glycine and glutamate, enters into the detoxification processes of endogenous products, such as peroxides which are the final pathway of many reactions caused by cardiovascular risk factors. It also acts on the exogenous compounds, such as pollutants, heavy metals and some drugs.

Changes in GSH homeostasis have been implicated in the etiology and progression of several diseases. A reduced bioavailability of GSH has been associated with neurodegenerative diseases such as Parkinson's and Alzheimer's or with increased risk of cardiovascular events.

The imbalance in the GSH homeostasis and aminothiols redox state is also involved in mechanisms that cause both chronic obstructive pulmonary and lung diseases and cystic fibrosis. Low levels of GSH have been found in individuals with HIV and are associated to reduced patients survival.

On the basis of previous data, it is conceivable that supplementation of GSH, whose concentrations decrease merely with age, may improve the endogenous antioxidant defense and may contribute to decrease of oxidants tissue damage, a typical characteristic of many acute and chronic diseases.

Several authors studied the effect of GSH oral administration in acute and in medium-long term treatment in healthy volunteers or in patients affected by different diseases. Unfortunately, they did not find any beneficial effect in terms of oxidative stress reduction and/or disease improvement. GSH was also administered intravenous, intramuscular or intrabronchial without positive results.

The efficacy of GSH treatment seems to be closely related to the degree of its absorption and to the increase of its concentrations in plasma and cells. Preliminary data obtained at the Institute of Clinical Physiology Institute of Milan in a small sample of healthy volunteers have shown that sublingual administration (100 mg) of a new preparation of L-glutathione (OXITION, PH&T S.r.l.) is able to increase over 4 h, plasma and erythrocyte GSH concentrations with an average of 70% compared to the endogenous physiological levels. This increase is not detectable after oral intake of the same molecule due to the gastrointestinal barrier. The primary objective of this study is to determine whether medium-term sublingual administration of reduced L-GSH for 4 weeks to male subjects with risk factor smoking habit and/or arterial hypertension results in improved endothelial function, as assessed by arterial FMD, when compared to placebo. A favourable response to study compound will result in a greater endothelium-dependent vasodilatory ability as assessed by the ratio between peak flow after reactive hyperaemia and basal flow. Secondary study objective is to determine differences between L-GSH supplementation and placebo in terms of oxidative stress markers.

Sixteen male healthy subjects will be randomized to sequential allocation to reduced L-GSH or placebo, according to the following inclusion criteria: age from 40 to 60 years, without any signs or symptoms of cardio-cerebro-vascular event at the enrolment, with smoking habit (>10 cigarette/die) and/or arterial hypertension (PAS≥140 mmHg and/or PAD≥90 mmHg or in anti-hypertensive treatment). Consenting subjects will be enrolled and sequentially assigned to study treatment following a double-blind, cross over, randomized and controlled experimental design (L-GSH versus placebo) with a 3-week wash-out period between the two treatments. Each intervention will last 4 weeks. Baseline evaluation includes interview for history and nutritional characterization, blood pressure and heart rate assessment, blood sampling for routine haematological analysis [serum fasting glucose (GLU), total cholesterol (TC), LDL cholesterol (LDL-C), HDL cholesterol (HDL-C), triglycerides (TG), creatinine (CREA), urea, gamma-glutamyl-transpeptidase (GGT), aspartate-amino transferase (AST) alanine-amino transferase (ALT)], and specific biochemical determination of endogenous redox status (total and reduced plasma aminothiols, total and reduced blood glutathione by HPLC) and oxidative stress mediators [plasma nitrotyrosine (NT), plasma malondialdehyde (MDA) and plasma 8-hydroxy-2'-deoxyguanosine (8-OHdG) by ELISA Kits]. FMD will be measured by a non invasive plethysmographic method (Endo-PAT2000) based on the registration of pulsatile blood volume in the fingertips of both hands.

After baseline assessment, patients will be randomized through a computer based procedure to active treatment or placebo in a 1:1 ratio. Study drug will be dispensed. At the 4-week follow-up, vital signs assessment, blood sampling for routine and specific biochemical determination, and FMD test will be again performed.

ELIGIBILITY:
Inclusion Criteria:

* informed consensus
* age from 40 to 60 years,
* without any signs or symptoms of cardio-cerebro-vascular event at the enrolment,
* smokers (>10 cigarette/die from almost 1 year)
* arterial hypertension (PAS≥140 mmHg and/or PAD≥90 mmHg or in anti-hypertensive treatment)

Exclusion Criteria:

* chronic assumption of acetylsalicylic acid and/or statins
* obesity defined as BMI ≥30 kg/m2
* diabetes mellitus defined as fasting glycemia >126 mg/dL
* dyslipidemia defined as LDL >155 mg/dL
* chronic renal dysfunction with Glomerular Filtration Rate<60 mL/min/1.73 m2
* in acetylcysteine treatment or with any other GSH-related molecules supplementation
* in vitamins supplementation or with other compounds derived from red rice (ARMOLIPID or similar).

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
endothelium-dependent vasodilation | Baseline and at 1 month after placebo or L-GSH treatment
  Registration of pulsatile blood volume in the fingertips of both hands will be assessed by a non invasive plethysmographic method (Endo-PAT2000, Itamar Medical Ltd., Caesarea, Israel) system. Endo-PAT device consists of two finger-mounted probes, which include a system of inflatable latex air-cushions within a rigid external case. The probe design allows the application of a constant and evenly distributed near-diastolic counterpressure within the entire probe, which increases sensitivity by unloading arterial wall tension, and prevents venous blood pooling to avoid venoarteriolar reflex vasoconstriction. Pulsatile volume changes of the fingertip are sensed by a pressure transducer and transferred to a personal computer where the signal is band pass-filtered (0.3 to 30 Hz), amplified, displayed, and stored.

SECONDARY OUTCOMES:
Oxidative stress markers | Baseline and at 1 month after placebo or L-GSH treatment
  Screening (V-1 - day -1): eligibility assessment; Baseline 1 (V0 - day 0): informed consent, interview, vital signs (blood pressure and heart rate), routine biochemistry (serum fasting glucose, total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, creatinine, urea, gamma-glutamyl-transpeptidase, aspartate-amino transferase, alanine-amino transferase), specific biochemistry (total and reduced blood glutathione, plasma nitrotyrosine, plasma malondialdehyde and plasma 8-hydroxy-2'-deoxyguanosine) flow-mediated dilation (FMD) assessment, randomization and dispense drug (L-GSH or placebo - 100 mg b.i.d.); Follow-up 1 (V1 - week 4): vital signs, routine biochemistry, specific biochemistry, FMD, adverse events; Baseline 2 (V2 - week 7/8): interview, vital signs, routine biochemistry, specific biochemistry, FMD and dispense drug (L-GSH or placebo - 100 mg b.i.d.); Follow-up 2 (V3 - week 11/12): vital signs, routine biochemistry, specific biochemistry, FMD, adverse events

OTHER OUTCOMES:
Adverse events | after 4, 8 and 12 weeks from the first visit V0
  The safety will be assessed by monitoring the adverse effects related with the administration of LGSH or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Jonica Campolo, MSc, Study Director — Insitute of Clinical Physiology CNR; Gianpalolo Micheloni, MD, Study Chair — Niguarda Ca' Granda Hospital
Locations (1):
- Oberdan Parodi, MD, Milan, Milan, Italy